CLINICAL TRIAL: NCT00003606
Title: Phase III Randomized Study of Cisplatin and Etoposide With or Without Epirubicin and Cyclophosphamide for Extensive Stage Small Cell Lung Cancer
Brief Title: Combination Chemotherapy in Treating Patients With Extensive Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000066683; FRE-FNCLCC-95012; EU-98021
Record Dates: First submitted 1999-11-01; First posted 2004-05-21 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Lung Cancer
Keywords: extensive stage small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Cisplatin; Cyclophosphamide; Epirubicin; Etoposide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: cisplatin
Drug: cyclophosphamide
Drug: epirubicin hydrochloride
Drug: etoposide
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. It is not yet known whether combination chemotherapy with or without epirubicin and cyclophosphamide is more effective in treating patients with extensive stage small cell lung cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of combination chemotherapy with or without epirubicin and cyclophosphamide in treating patients who have extensive stage small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the overall survival and survival without recurrence of patients with extensive stage small cell lung cancer after receiving cisplatin and etoposide with or without epirubicin and cyclophosphamide. II. Compare the relative dose and intensity of cisplatin and etoposide between the two groups of patients. III. Compare the complete and objective response rate and quality of life of these patients. IV. Compare the toxic effects of these 2 regimens in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to one of two treatment arms. Arm I: Patients receive etoposide IV on days 1 and 3 and cisplatin IV on day 2. Arm II: Patients receive etoposide and cisplatin as in arm I, plus epirubicin IV on day 1 and cyclophosphamide IV on days 1 and 3. Treatment is repeated in both arms every 28 days for up to 6 courses. Patients who achieve a partial or complete response receive cerebral and/or thoracic radiotherapy. Patients with residual tumor may receive oral etoposide for 3 of every 4 weeks. Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 216 patients will be accrued for this study within 2.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven extensive stage small cell lung cancer Extends beyond hemithorax and supraclavicular lymph nodes Pleural effusions allowed Bidimensionally measurable disease Bone marrow metastases allowed No symptomatic CNS metastases or carcinomatous meningitis

PATIENT CHARACTERISTICS: Age: 18 to 75 Performance status: 0-2 Life expectancy: Not specified Hematopoietic: Neutrophil count at least 2,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 times normal Renal: Creatinine less than 1.24 mg/dL OR Creatinine clearance greater than 60 mL/min Cardiovascular: No cardiac insufficiency No uncontrolled cardiac disease LVEF greater than 50% OR ECHO greater than 30% Other: Not pregnant Fertile patients must use effective contraception No psychoses No active infection No loss of weight greater than 10% during the last 3 months No other malignancy except nonmelanomatous skin cancer or stage I cervical cancer

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior or concurrent immunotherapy Chemotherapy: No prior or other concurrent chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior or concurrent radiotherapy Surgery: No prior or concurrent surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 1996-03 (Actual); Primary Completion 1999-10-01 (Actual); Study Completion 2001-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Louis Pujol, MD, Study Chair — Hopital Arnaud de Villeneuve
Locations (1):
- Hopital Arnaud de Villeneuve, Montpellier, France

REFERENCES:
- [Result] Pujol JL, Daures JP, Riviere A, Quoix E, Westeel V, Quantin X, Breton JL, Lemarie E, Poudenx M, Milleron B, Moro D, Debieuvre D, Le Chevalier T. Etoposide plus cisplatin with or without the combination of 4'-epidoxorubicin plus cyclophosphamide in treatment of extensive small-cell lung cancer: a French Federation of Cancer Institutes multicenter phase III randomized study. J Natl Cancer Inst. 2001 Feb 21;93(4):300-8. doi: 10.1093/jnci/93.4.300. PMID 11181777
- [Result] Pujol JL, Duares JP, Riviere A, et al.: Doublet etoposide - cisplatin (EP) versus quadruplet cisplatin - cyclophosphamide - epirubicin - etoposide (PCDE) in extensive disease small cell lung cancer (Ed-SCLC): a FNCLCC phase III multicenter study. [Abstract] Proceedings of the American Society of Clinical Oncology 19: A-1892, 2000.